CLINICAL TRIAL: NCT06801730
Title: Exploratory Study of Irinotecan Liposomes Combined With Bevacizumab in the Treatment of Progressive or Recurrent Glioma
Brief Title: Irinotecan Liposomes Combined With Bevacizumab in the Treatment of Recurrent Glioma
Acronym: NALIRIBVRG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhifeng Tian,MD (Other)
Responsible Party: Sponsor-Investigator, Zhifeng Tian,MD, Head and neck esophageal Center, The Central Hospital of Lishui City
Organization: The Central Hospital of Lishui City (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024(I)-107-01
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Glioma
Keywords: Irinotecan liposomes; Bevacizumab; Recurrent; Glioma
MeSH Terms: conditions — Glioma; Recurrence | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Single-arm prospective exploratory study
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome combined with bevacizumab (Experimental): Irinotecan liposomes, 50mg/m2, d1, 90 min intravenously, Q2W; Bevacizumab 10mg/kg, d1, Q2W;
  Interventions: Drug: Irinotecan liposome combined with bevacizumab

INTERVENTIONS:
Drug: Irinotecan liposome combined with bevacizumab — Irinotecan liposomes, 50mg/m2, d1, 90 min intravenously, Q2W; Bevacizumab 10mg/kg, d1, Q2W;

SUMMARY:
With the optimization of the dosage form of irinotecan, the replacement of ordinary irinotecan with irinotecan liposomes should improve the safety and the expected efficacy. Therefore, an exploratory study on the treatment progress of irinotecan liposomes combined with bevacizumab for recurrent brain glioma should be conducted. To evaluate the efficacy and safety of irinotecan liposomes combined with bevacizumab in the treatment of progressive/recurrent brain glioma, so as to provide more treatment options for patients with brain glioma.

DETAILED DESCRIPTION:
This study was to observe the efficacy and safety of irinotecan liposomes combined with bevacizumab in the treatment of progressive/recurrent brain glioma. The study was a single-center, single-arm, prospective study. Patients with progressive/recurrent glioma who met the inclusion criteria and did not meet the exclusion criteria were treated with irinotecan liposome combined with beizumab. The optimal ORR of patients during treatment was mainly evaluated, and the DCR, DoR, PFS, OS, and safety of patients were mainly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old;
* Patients diagnosed with glioma by histology, patients with progress in first-line therapy, including postoperative recurrence, progress in first-line standard therapy, and patients unable to undergo surgery/radiotherapy;
* no previous treatment with irinotecan or irinotecan liposomes;
* At least one measurable or evaluable lesion according to RANO criteria;
* ECOG score is 0~1;
* Good bone marrow and organ function: ① Neutrophils (ANC) ≥1.5×109/L, platelets (PLT) ≥100×109/L, hemoglobin (Hb) ≥90g/L, white blood cells (WBC) ≥3.0×109/L, albumin (ALB) ≥32 g/L, and no bleeding tendency; ② AST, ALT and alkaline phosphatase (ALP) were all ≤2.5× upper limit of normal range (ULN), and ≤5×ULN when liver metastases occurred; Total bilirubin ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated according to Cockroft-Gault);
* Expected survival ≥3 months;
* Can understand the situation of this study, patients and (or) legal representatives voluntarily agree to participate in this study and sign informed consen;

Exclusion Criteria:

* Patients allergic to the investigational drug and its excipients;
* Known or suspected central nervous system metastasis;
* The use of potent depressants or inducers of CYP3A, CYP2C8, and UGT1A1 (anticonvulsants [phenytoin, phenobarbital, or carbamazepine], rifampicin, rifambutin, St.John's.) could not be discontinued or were not discontinued within 2 weeks prior to enrollment Wort], grapefruit juice, clarithromycin, itraconazole, Lopinavir, Nefazodone, Nelfinavir, Ritonavir, Saquinavir, Terrapivir, voriconazole, Azanavir, Gefilozil, indinavir, etc.);
* There are signs and symptoms of intestinal obstruction;
* have had other malignant tumors within the past 5 years or currently, except for cured cervical carcinoma in situ, uterine carcinoma in situ and non-melanoma skin cancer;
* Pregnant or lactating female patients, patients of childbearing age who refuse to accept contraceptive measures;
* Patients considered by the investigator to be unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of randomization until the date of one year
  The proportion of patients with optimal tumor response, complete response (CR) or partial response (PR) assessed based on the RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The time from the start of treatment to the first recording of PD or death, whichever occurs first
Overall survival | From date of randomization until the date of death from any cause, assessed up to 24 months
  The time between the start of treatment and the first recorded death

CONTACTS AND LOCATIONS:
Overall Officials: Zhifeng Tian, Study Chair — The Central Hospital of Lishui City
Locations (1):
- The central Hospital of Lishui City, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
At the end of the test, the decision is made according to the test results